CLINICAL TRIAL: NCT05479695
Title: The Effect of Insoles on Functional Capacity, Quality of Life, Balance and Plantar Pressure in Patient With Adolescent Idiopathic Scoliosis Using Chêneau Type Spinal Orthosis
Brief Title: The Effect Insoles on Functional Capacity With Adolescent Idiopathic Scoliosis Using Spinal Orthosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, merve arslan, Research Assistant, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: mervearslan
Record Dates: First submitted 2021-03-12; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Scoliosis; Adolescence; Pressure Area; Scoliosis; Orthosis
Keywords: Adolescent Idiopathic Scoliosis; Scoliosis Brace; Insoles
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Intervention Model Description: The first group uses spinal orthoses. The second group uses spinal orthosis and insoles.
Who Masked: Participant
Masking Description: 54 pre-filled sealed envelopes were prepared for the randomization process of the participants who met the inclusion and exclusion criteria determined in the study. 27 envelope series consists of 1 number and 27 envelope series consists of 2 number. The control group (KG) using Chêneau type spinal orthosis was given number 1, and the group using Chêneau type spinal orthosis and insoles (TG) was given number 2. Each of the participants chose one of the sealed envelopes in turn. Participants included in the study were randomly assigned to the KG group or the TG group according to the number on the selected envelope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient who use spinal orthoses and insoles (Experimental): Spinal Orthoses: Devices that used in spinal deformities. Insoles: Devices that used in foot deformities.
  Interventions: Device: Spinal Orthoses and Insoles
- Patient who use only spinal orthoses (Other): Spinal Orthoses: Devices that used in spinal deformities.
  Interventions: Device: Spinal Orthoses

INTERVENTIONS:
Device: Spinal Orthoses and Insoles — Evaluation of scoliosis treatment in people using spinal orthoses and insoles
  Arms: Patient who use spinal orthoses and insoles
Device: Spinal Orthoses — Evaluation of scoliosis treatment in people using spinal orthoses
  Arms: Patient who use only spinal orthoses

SUMMARY:
Adolescent Idiopathic Scoliosis; by problem of stabilty causes postural changes, because of this reason patient with scoliosis needs to assesment by risk of balance. Postural adjustments are required, both in a static stance and during walking. Insoles from foot orthoses support better postural balance and control.

It has been reported that approximately 87% of scoliosis patients have pelvic asymmetry, and patients with scoliosis with a Cobb angle of 15⁰ or more have balance problems in their feet. Foot orthoses (FO) correct pelvic asymmetry and reduce lower extremity joint angles during walking.

In the literature, although there are studies such as balance assessment and plantar pressure analysis in Adolescent Idiopathic Scoliosis (AIS) patients, there are not enough studies on the effect of insoles used in scoliosis patients, and it has been observed that there is no study on the effect of insoles on treatment in patients using spinal orthosis.

The aim of this study is to investigate the effect of insoles on the treatment of scoliosis patients using Chêneau type spinal orthosis.

In the study; The effect of insoles on patients with 20-45⁰ curvature, adolescent idiopathic scoliosis and using Chêneau type spinal orthosis; It was planned to investigate the groups using and not using insoles at the beginning of the treatment and after 3 months of follow-up by comparing the results of Cobb angle measurement, functional capacity assessment test, quality of life assessment test, balance test and plantar pressure analysis.

DETAILED DESCRIPTION:
Adolescent Idiopathic Scoliosis (AIS) is a three-dimensional deformity of the spine that is commonly seen in individuals aged 10-19 years, and spinal orthosis application, one of the conservative treatment methods, is widely preferred today. Spinal orthosis application in individuals with scoliosis may adversely affect functional capacity, quality of life, balance and plantar pressure. The aim of this study is to determine the use of insoles for 3 months in AIS individuals using Chêneau type spinal orthosis functional capacity, quality of life, balance and the effect of plantar pressure is to investigate. Study group included 42 individuals aged between 10-19 with a Cobb angle of 20-45⁰. Participants were randomly separated into 2 groups; Control-KG (n=21) and using insoles-TG (n=21). While only Chêneau type spinal orthosis was applied to KG group for 3 months, Chêneau type spinal orthosis and insoles were applied to TG group. Measurements were repeated after one week of spinal orthosis application and at the end of the 3rd month. The 6 Minute Walk Test (6 MWT) was used to evaluate the functional capacity of the participants, the Scoliosis Research Society-22 (SRS-22) for quality of life, and the Sensor Medica Maxi pedobarographic device for balance and plantar pressure measurements.

ELIGIBILITY:
Inclusion criteria;

* Adolescent idiopathic scoliosis patients between the ages of 10-19
* Cobb angle to be in the range of 20-45 °
* Adolescent idiopathic scoliosis patients who will use Chêneau type spinal orthosis for the first time or who will be renewed with a Chêneau type spinal orthosis
* Absence of neurological problems
* Differences in plantar pressure analysis of the two lower extremities

Exclusion criteria;

* Previously used insoles
* Finding a neurological problem
* Those with congenital lower extremity deformities
* Patients with lower extremity length difference more than 2 cm

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2021-05-22 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
6-minute walk test | Change from Baseline of treatment at 3 months
  assessment of functional capacity
Scoliosis Research Society (SRS-22 test) | Change from Baseline of treatment at 3 months
  assessment of quality of life
sway balance test | Change from Baseline of treatment at 3 months
  assessment of postural balance
plantar pressure analysis | Change from Baseline of treatment at 3 months
  static and dynamic plantar pressure analysis

CONTACTS AND LOCATIONS:
Overall Officials: Sena OZDEMİR GORGU, Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No